CLINICAL TRIAL: NCT05197231
Title: Investigating the Anabolic Response to Resistance Exercise During Critical Illness: The ARTIST-1 Randomized Controlled Trial
Brief Title: Investigating the Anabolic Response to Resistance Exercise During Critical Illness
Acronym: ARTIST-1
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical barriers to recruitment.
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Martin Sundstrom Rehal, Principal Investigator, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K 2021-10530
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Critical Illness; Muscle Loss
Keywords: Physiotherapy; Resistance exercise; Amino acids; Muscle protein balance
MeSH Terms: conditions — Critical Illness; Muscular Atrophy | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV amino acids + standardized physiotherapy with lower limb resistance exercise. (Experimental): Research subjects randomized to the intervention group will receive an infusion of IV amino acids during a session of protocolized physiotherapy that includes a knee extension resistance exercise targeting the thigh muscles. The supplemental amino acid infusion will continue up until 90 minutes after the subject has returned to bed rest.
  Interventions: Procedure: Resisted knee extension exercise; Drug: IV amino acids
- IV amino acids + standardized physiotherapy. (Active Comparator): Research subjects randomized to the control group will receive an infusion of IV amino acids during a session of protocolized physiotherapy NOT including lower limb resistance exercise. The supplemental amino acid infusion will continue up until 90 minutes after the subject has returned to bed rest.
  Interventions: Drug: IV amino acids

INTERVENTIONS:
Procedure: Resisted knee extension exercise — Patients in the intervention group will perform a seated knee extension exercise in three sets. Resistance will be adjusted using ankle weights, targeting 8-12 repetitions per set.
  Arms: IV amino acids + standardized physiotherapy with lower limb resistance exercise.
Drug: IV amino acids — IV amino acids (Glavamin, Fresenius Kabi) delivered by continuous infusion at a rate of 0.1 g/kg/h. The infusion is started immediately prior to physiotherapy and continued until all blood samples required for outcome assessment are collected during a 90-minute resting period after the exercise session.
  Other Names: Glavamin (Fresenius Kabi)

SUMMARY:
ICU patients often suffer from rapid and severe muscle loss. It is not known if physical therapy can mitigate the muscle wasting associated with critical illness.

The aim of this study is to investigate the effects of resistance exercise on muscle protein turnover in ICU patients. The investigators hypothesize that resistance exercise, in addition to amino acid supplementation and routine physiotherapy, results in an improved lower limb muscle protein balance compared to amino acid supplementation and routine physiotherapy alone.

DETAILED DESCRIPTION:
Background

The debilitating impact of critical illness has been recognized for several decades. Disability related to intensive care is now described as a syndrome called ICU-acquired weakness (ICUAW). ICUAW affects up to 70% of ICU patients and is most common with higher illness severity. Patients that develop ICUAW require longer hospitalization and have a higher risk of death. Weakness also has significant long-term consequences, and is associated with significant health care costs, delayed return to work, and overall poor quality of life.

Preventing or reducing muscle atrophy is a potential way to counteract weakness. Critical illness is associated with a rapid loss of skeletal muscle. Studies in exercise physiology have demonstrated that resistance training and amino acid ingestion have synergistic effects on muscle protein synthesis in healthy subjects. It is therefore an appealing therapy to counteract muscle wasting in the ICU.

Despite several clinical trials, there is equipoise regarding the efficacy of exercise in improving physical function in-ICU or after discharge. These mixed signals are unsurprising given the heterogeneous causes of ICUAW. Only a few studies in this field assess muscle architecture or cellular signaling in response to training. However, the gold standard in determining the anabolic response to exercise is to directly measure the effect on protein synthesis and breakdown. To our knowledge there is still no published research using this methodology to assess the effects of exercise interventions in critically ill patients.

Aim and hypothesis

The overall aim of this project is to determine the anabolic response to resistance exercise during critical illness. The investigators hypothesize that resistance exercise, in addition to amino acid supplementation and routine physiotherapy, results in an improved muscle protein balance in ICU patients compared to amino acid supplementation and routine physiotherapy alone (primary outcome). The effect of the intervention on other parameters of muscle protein kinetics and within-group differences in protein kinetics before and after physiotherapy will be assessed as secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years) patient admitted to the ICU of the study site.
2. Patient deemed suitable for active mobilization by the attending physician and physiotherapist.
3. Not expected to be discharged or transferred from the unit within 24 h of enrollment.
4. Functioning arterial catheter in situ.

Exclusion Criteria:

1. Not able to provide informed consent.
2. Systemic anticoagulation with LMWH/UFH/DOAC in therapeutic dose range for deep vein thrombosis or pulmonary embolism, or dual antiplatelet therapy. If LMWH is administered twice daily, the patient is eligible for participation provided that vascular access is performed at nadir prior to the first daily dose.
3. Clinically significant inherited or acquired disorder of hemostasis.
4. Morbid obesity that interferes with femoral cannulation or doppler measurements.
5. Hemodynamic instability requiring ongoing volume resuscitation with crystalloid solutions or blood products.
6. Lower-limb amputee.
7. Lower-limb artherosclerotic disease with critical ischemia.
8. Metastatic cancer or active hematological malignancy.
9. Inherited disorder of amino acid metabolism.
10. Chronic muscle, neuromuscular and neurologic disease with prior documentation of clinically significant lower-limb involvement.
11. Pregnancy.
12. CAM-ICU screening positive for delirium.
13. Single organ failure not requiring invasive mechanical ventilation prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in change in lower limb protein balance | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The difference between the experimental and active comparator group in change in lower limb protein balance (nmol Phenylalanine/min) from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.

SECONDARY OUTCOMES:
Between-group difference in change in lower limb protein synthesis | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The difference between the experimental and active comparator group in change in lower limb protein synthesis (nmol Phenylalanine/min) from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.
Between-group difference in change in lower limb protein breakdown | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The difference between the experimental and active comparator group in change in lower limb protein breakdown (nmol Phenylalanine/min) from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.
Between-group difference in change in lower limb 3-methylhistidine rate of appearance | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The difference between the experimental and active comparator group in change in lower limb 3-methylhistidine rate of appearance (nmol 3-methylhistidine/min) from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.
Within-group change in lower limb protein balance (experimental group) | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The change in lower limb protein balance (nmol Phenylalanine/min) in the experimental group, from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.
Within-group change in lower limb protein balance (active comparator group) | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The change in lower limb protein balance (nmol Phenylalanine/min) in the active comparator group, from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.
Within-group change in lower limb protein synthesis (experimental group) | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The change in lower limb protein synthesis (nmol Phenylalanine/min) in the experimental group, from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.
Within-group change in lower limb protein synthesis (active comparator group) | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The change in lower limb protein synthesis (nmol Phenylalanine/min) in the active comparator group, from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.
Within-group change in lower limb protein breakdown (experimental group) | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The change in lower limb protein breakdown (nmol Phenylalanine/min) in the experimental group, from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.
Within-group change in lower limb protein breakdown (active comparator group) | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The change in lower limb protein breakdown (nmol Phenylalanine/min) in the active comparator group, from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.
Within-group change in lower limb 3-methylhistidine rate of appearance (experimental group) | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The change in lower limb 3-methylhistidine rate of appearance (nmol 3-methylhistidine/min) in the experimental group, from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.
Within-group change in lower limb 3-methylhistidine rate of appearance (active comparator group) | Time = 165-180 minutes from start of study protocol to approximate Time = 315 minutes from start of study protocol.
  The change in lower limb 3-methylhistidine rate of appearance (nmol 3-methylhistidine/min) in the active comparator group, from baseline to post-physiotherapy. Blood samples and lower limb blood flow measurements to determine protein kinetics are performed at baseline (before IV amino acids and physiotherapy) and at 30, 60, and 90 minutes during bed rest after the physiotherapy session.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sundström Rehal, MD PhD, Principal Investigator — Karolinska University Hospital; Olav Rooyackers, PhD, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batt J, Herridge MS, Dos Santos CC. From skeletal muscle weakness to functional outcomes following critical illness: a translational biology perspective. Thorax. 2019 Nov;74(11):1091-1098. doi: 10.1136/thoraxjnl-2016-208312. Epub 2019 Aug 20. PMID 31431489
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Plank LD, Connolly AB, Hill GL. Sequential changes in the metabolic response in severely septic patients during the first 23 days after the onset of peritonitis. Ann Surg. 1998 Aug;228(2):146-58. doi: 10.1097/00000658-199808000-00002. PMID 9712558
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Wolfe RR. Skeletal muscle protein metabolism and resistance exercise. J Nutr. 2006 Feb;136(2):525S-528S. doi: 10.1093/jn/136.2.525S. PMID 16424140
- [Background] Doiron KA, Hoffmann TC, Beller EM. Early intervention (mobilization or active exercise) for critically ill adults in the intensive care unit. Cochrane Database Syst Rev. 2018 Mar 27;3(3):CD010754. doi: 10.1002/14651858.CD010754.pub2. PMID 29582429
- [Background] Connolly B, Salisbury L, O'Neill B, Geneen L, Douiri A, Grocott MP, Hart N, Walsh TS, Blackwood B; ERACIP Group. Exercise rehabilitation following intensive care unit discharge for recovery from critical illness. Cochrane Database Syst Rev. 2015 Jun 22;2015(6):CD008632. doi: 10.1002/14651858.CD008632.pub2. PMID 26098746
- [Background] Fossat G, Baudin F, Courtes L, Bobet S, Dupont A, Bretagnol A, Benzekri-Lefevre D, Kamel T, Muller G, Bercault N, Barbier F, Runge I, Nay MA, Skarzynski M, Mathonnet A, Boulain T. Effect of In-Bed Leg Cycling and Electrical Stimulation of the Quadriceps on Global Muscle Strength in Critically Ill Adults: A Randomized Clinical Trial. JAMA. 2018 Jul 24;320(4):368-378. doi: 10.1001/jama.2018.9592. PMID 30043066
- [Background] Hickmann CE, Castanares-Zapatero D, Deldicque L, Van den Bergh P, Caty G, Robert A, Roeseler J, Francaux M, Laterre PF. Impact of Very Early Physical Therapy During Septic Shock on Skeletal Muscle: A Randomized Controlled Trial. Crit Care Med. 2018 Sep;46(9):1436-1443. doi: 10.1097/CCM.0000000000003263. PMID 29957714

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT05197231/Prot_SAP_000.pdf